CLINICAL TRIAL: NCT06836453
Title: Evaluation of New System for β-adrenergic Sweat Test in the Context of Stratification of Patient With Cystic Fibrosis
Brief Title: Evaluation of New Device for Beta-adrenergic Sweat Test in the Context of Stratification of Patient With Cystic Fibrosis
Acronym: BESTRACYFIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIV-24-02-046176
Record Dates: First submitted 2025-01-06; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Beta-adrenergic sweat test; Stratification
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EVALUATION OF NEW SYSTEM FOR β-ADRENERGIC SWEAT TEST IN THE CONTEXT OF STRATIFICATION OF PATIENT WI (Experimental): First session (50 minutes):
  1. Left arm: Iontophoresis using the Macroduct for the cholinergic and β-adrenergic stimulation (2 iontophoresis), then bubble test.
  2. right arm: Iontophoresis using the Macroduct for the cholinergic and β-adrenergic stimulation (2 iontophoresis), then evaporimetry.
  Second session (50 minutes):
  1. Left arm: Iontophoresis using the Macroduct for the cholinergic and intradermal injection for the β-adrenergic stimulation, then bubble test.
  2. Right arm: Iontophoresis using the Macroduct for the cholinergic and intradermal injection for the β-adrenergic stimulation, then evaporimetry.
  Interventions: Device: Sweat stimulation and secretion quantification

INTERVENTIONS:
Device: Sweat stimulation and secretion quantification — First session (50 minutes): a. Left arm: Iontophoresis using the Macroduct for the cholinergic and β-adrenergic stimulation (2 iontophoresis), then bubble test. b. right arm: Iontophoresis using the Macroduct for the cholinergic and β-adrenergic stimulation (2 iontophoresis), then evaporimetry.
  Second session (50 minutes): a. Left arm: Iontophoresis using the Macroduct for the cholinergic and intradermal injection for the β-adrenergic stimulation, then bubble test. b. Right arm: Iontophoresis using the Macroduct for the cholinergic and intradermal injection for the β-adrenergic stimulation, then evaporimetry.

SUMMARY:
This is a clinical study to evaluate a new medical system used to perform a sweat secretion-based test for the diagnosis of cystic fibrosis.

This clinical study will involve around 150 individuals in Belgium, including 50 healthy individuals, 50 carriers and 50 patients with cystic fibrosis.

The primary objective is to implement a new system for diagnosing cystic fibrosis according to their response to the beta-adrenergic test.

First session (50 minutes):

1. Left arm: Iontophoresis using the Macroduct for the cholinergic and β-adrenergic stimulation (2 iontophoresis), then bubble test.
2. right arm: Iontophoresis using the Macroduct for the cholinergic and β-adrenergic stimulation (2 iontophoresis), then evaporimetry.

Second session (50 minutes):

1. Left arm: Iontophoresis using the Macroduct for the cholinergic and intradermal injection for the beta-adrenergic stimulation, then bubble test.
2. Right arm: Iontophoresis using the Macroduct for the cholinergic and intradermal injection for the beta-adrenergic stimulation, then evaporimetry.

The secondary objectives of this clinical research are:

* Determining the best mode of administration for beta-adrenergic stimulation
* Assessing the best quantification of sweat secretion
* Comparing the response of the control group and the carrier group
* Evaluating the stratification of people with cystic fibrosis according to CFTR dysfunction

The test consists of 5 steps:

1. sweat stimulation by cholinergic pathway
2. sweat secretion quantification
3. cystic fibrosis specific stimulation: beta-adrenergic pathway
4. sweat secretion quantification
5. analysis Both techniques of sweat stimulation and secretion quantification will be performed and compared to each other. Each participants will therefore have 2 sessions on both arms, with a minimum of one hour between the two sessions.

At each stimulation steps (step 1 to 3), the pain level during the test will be evaluated by self assessment in adults with Visual Analog Scale and children 2 to 6 years old with Faces Pain Scale - Revised or a hetero-assessment of pain for children less than 2 years old with douleur aigue du nouveau-ne scale.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a rare genetic disease affecting 1 baby in 2,850 live births in Belgium and associated with high morbidity and mortality. CF is caused by CFTR mutations resulting in loss-of-function of the CFTR protein. It leads to dramatic abnormalities in transepithelial ion transport and the production of thick mucus obstructing airways and duct lumens of exocrine glands. The gold standard for CF diagnosis is an accurate Gibson and Cooke sweat test which is very sensitive to lost or abrogated CFTR function, but shows a logarithmic relationship between sweat Cl - content and CFTR function: e.g. a 5% residual CFTR function is associated with sweat Cl- concentrations found below the diagnostic threshold (<60 mmol/L). Consequently, diagnosing CF is challenging in borderline cases and/or in the presence of CFTR mutations not recognized as disease-causing (CFTR2 data base; https://cftr2.org/). Contrary to routine sweat test measuring the CFTR-mediated reabsorption of Cl- in the sweat duct, beta-adrenergic sweat secretion test (BAST) measures CFTR mediated secretion of Cl- in the secretory coil of the sweat gland . Sato and Sato discovered in the early 1980s that CFTR-mediated sweat secretion can be stimulated with β-adrenergic agonists if the thermoregulative cholinergic sweat secretion is simultaneously inhibited with atropine . β-adrenergic sweat secretion was absent in people with CF (pwCF) and half-maximal in healthy heterozygous carriers of CFTR mutation (HTZ). Therefore, BAST seems to be a highly sensitive CFTR bioassay suitable for screening of CFTR dysfunction, monitoring the efficacy of new therapeutic interventions and differential diagnosis of exocrine pancreatic sufficient-CF, CFTR-Related disease and cystic fibrosis screen positive and finallyinconclusive diagnosis. BAST detect the relative improvement due to a novel treatment, while at the same time show that the levels did not return to a normal range. The available measurement range can thus be used to assess the individual response to therapeutic interventions, but can also be used to stratify patients in the intermediate range of activity, which fall into a spectrum, ranging from a severe loss of function in classical cystic fibrosis to the cystic fibrosis related disease with a relatively lowered activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* carriers (e.g. parents of people with cystic fibrosis)
* people with known cystic fibrosis or classified as cystic fibrosis related disease

Exclusion Criteria:

* Any individual with skin lesions affecting the measurement site
* pregnant or breastfeeding women
* participants with temporary or definitive disabilities to give consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Sweat secretion | 2 hours
  To distinguish people with cystic fibrosis, the beta-adrenergic sweat rate less than or equal to 4.5 TEWL and the beta-adrenergic:cholinergic ratio less than or equal to 0.05 measured by the evaporimetry test will be used.
  For the bubble test, a β-adrenergic sweat rate of less than 0.16 nL/min will be used to define a CF base range.

SECONDARY OUTCOMES:
Pain assessment score | 2 hours
  Pain during the test will be assessed by self-report in adults and children >6 years old, or by hetero-report in children <6 years old. A score > 3-4/10 leads to discontinuation of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Gohy, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Background] Pallenberg ST, Junge S, Ringshausen FC, Sauer-Heilborn A, Hansen G, Dittrich AM, Tummler B, Nietert M. CFTR modulation with elexacaftor-tezacaftor-ivacaftor in people with cystic fibrosis assessed by the beta-adrenergic sweat rate assay. J Cyst Fibros. 2022 May;21(3):442-447. doi: 10.1016/j.jcf.2021.10.005. Epub 2021 Oct 29. PMID 34756683
- [Background] Zampoli M, Verstraete J, Nguyen-Khoa T, Sermet-Gaudelus I, Zar HJ, Gonska T, Morrow BM. beta-adrenergic sweat test in children with inconclusive cystic fibrosis diagnosis: Do we need new reference ranges? Pediatr Pulmonol. 2023 Jan;58(1):187-196. doi: 10.1002/ppul.26179. Epub 2022 Oct 17. PMID 36193559
- [Background] Reynaerts A, Vermeulen F, Mottais A, Gohy S, Lebecque P, Frederick R, Vanbever R, Leal T. Needle-free iontophoresis-driven beta-adrenergic sweat rate test. J Cyst Fibros. 2022 May;21(3):407-415. doi: 10.1016/j.jcf.2021.08.012. Epub 2021 Sep 4. PMID 34489187